CLINICAL TRIAL: NCT06881667
Title: US Development and Evaluation Study of a Patch-Based PSG System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Onera BV (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CIP_Protocol_Onera_D01
Record Dates: First submitted 2025-02-26; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Sleep Disorder (Disorder)
Keywords: sleep disordered breathing; sdb; sleep apnea; obstructive sleep apnea; apnea; home PSG; PSG; PSG type 2; PSG type II; sleep diagnostics; home
MeSH Terms: conditions — Sleep Wake Disorders; Sleep Apnea Syndromes; Sleep Apnea, Obstructive; Apnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Home PSG Assessment (Experimental): Testing of the Onera STS in the home environment with the current device shipment method and instructions.
  Interventions: Device: Home PSG Assessment

INTERVENTIONS:
Device: Home PSG Assessment — Testing of the Onera STS in the home environment with the current device shipment method and instructions.

SUMMARY:
The purpose of this study is continue the development and evaluation of the Onera system as well as the procedures and best practices for dispensing, instruction, use and reportability of results.

DETAILED DESCRIPTION:
The diagnostic gold standard to detect a sleep disorder in the presence of a comorbidity is attended, inpatient, polysomnography (PSG)1. Currently, these tests are limited to the in-patient setting in the sleep laboratory, which requires a large number of personnel, and the PSG studies are time-consuming and expensive to conduct. PSG studies are also burdensome for patients, as they require each patient to sleep at the hospital for at least one night while wearing multiple electrodes and other physiological monitoring equipment attached to the head, face, torso, and legs, which makes sleeping difficult and limits movement. A portable PSG device that does not incorporate traditional leads and electrodes would facilitate sleep studies and allow such studies to be done in other locations and be performed more quickly and easily. Studies outside the hospital setting using an optimized, portable PSG device would be easier for sleep technicians to set up and allow each patient to sleep more comfortably.

Onera STS is a wearable system for measuring physiological signals during a PSG study that was designed to overcome the limitations described above that are associated with attended, inpatient PSG. The Onera STS performs electroencephalography (EEG), electrooculography (EOG), electromyography (EMG), and electrocardiography (ECG) and also measures respiratory signals, nasal pressure, oxygen saturation, activity, body position, and snoring loudness via four sensor patches applied to the forehead, upper chest, abdomen, and lower leg. These sensor patches eliminate the need for individual leads and separate electrodes. When used in an in-patient setting, setup time can be reduced compared to the classical PSG setup. The Onera STS system is FDA approved (510k) for the purpose of monitoring physiological parameters intended to provide information which is used to take decisions on the diagnosis of sleep disorders.

The purpose of this study is continue the development and evaluation of the Onera system as well as the procedures and best practices for dispensing, instruction, use and reportability of results.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Referral for a suspected sleep disorder requiring a sleep diagnostic study

Exclusion Criteria:

* Inability to provide informed consent
* History of allergic reactions to adhesives or hydrogels or a family history of adhesive skin allergies
* Severe skin condition at sites of patch administration such as wounds, burns or on any damaged skin
* Has an implanted cardiac stimulator or diaphragmatic pacer
* Has an anatomical abnormality that, in the opinion of the Principal Investigator, makes the subject ineligible for inclusion
* Will be exposed to high-frequency surgical equipment, near strong magnetic fields or with devices such as MRIs, external cardiac stimulators during their use of the Onera device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-08-04 (Actual); Primary Completion 2024-09-02 (Actual); Study Completion 2024-09-02 (Actual)

PRIMARY OUTCOMES:
Study Success Rate | Assessment will be completed within one month after completion of the sleep study.
  Number of studies and reports scored to the AASM Scoring Manual version 2.6, 2020 considered acceptable for clinical use by the lead clinician on the study. A successful sleep study that can be used for diagnostic purposes indicates that the device application and signal collection was successful to assess device feasibility.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - The Sleep Disorders Center of Alabama, Birmingham, Alabama
  - Clayton Sleep Institute, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No
Commercially Sensitive

REFERENCES:
- [Derived] Uhles M, Alisic S, Brown A, Doekel R, Booth W, Ojile J. Feasibility and acceptance of self-applied home type-II PSG studies with a patch-based device. Sleep Breath. 2025 Oct 28;29(6):336. doi: 10.1007/s11325-025-03503-z. PMID 41148462